CLINICAL TRIAL: NCT01370044
Title: Carbon Dioxide (Carbogen) for the Treatment of Febrile Seizures
Acronym: CARDIF
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: results of interim analysis (not safety relevant)
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Markus Schuelke, M.D., Prof. Dr. med. Markus Schuelke, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CARDIF
Record Dates: First submitted 2011-05-20; First posted 2011-06-09 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Febrile Seizure
Keywords: Febrile Seizure; Carbon Dioxide; Carbogen; Respiratory Alkalosis
MeSH Terms: conditions — Seizures, Febrile; Alkalosis, Respiratory | interventions — carbogen; Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Verum (Experimental): Verum arm receiving Carbogen
  Interventions: Drug: Carbogen
- Placebo (Placebo Comparator): Placebo arm receiving oxygen
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carbogen — 3 minutes administration of carbogen
  Other Names: Low pressure flask with mask containing 6 L carbogen
  Arms: Verum
Drug: Placebo — 3 minutes administration of oxygen
  Other Names: Low pressure flask with mask containing 6 L oxygen
  Arms: Placebo

SUMMARY:
The aim of this clinical trail is to evaluate the efficacy of a Carbogen inhalation in patients with febrile seizures compared to a placebo-inhalation.

Further aims are the evaluation of the safety of the Carbogen inhalation via a low-pressure can with a breathing mask in a home-setting, the manageability of the Carbogen inhalation via a low pressure can with a breathing mask in a home-setting or on the way (mobility), the quality of life of the parents and children using the low pressure can with a breathing mask in a home-setting or on the way (mobility) and the contentment and anxiety of the parents.

DETAILED DESCRIPTION:
For detailed protocol see:

Ohlraun S, Wollersheim T, Weiß C, Martus P, Weber-Carstens S, Schmitz D, Schuelke M. CARbon DIoxide for the treatment of Febrile seizures: rationale, feasibility, and design of the CARDIF-study. J Transl Med. 2013 Jun 27;11:157. doi: 10.1186/1479-5876-11-157.

BACKGROUND: 2-8% of all children aged between 6 months and 5 years have febrile seizures. Often these seizures cease spontaneously, however depending on different national guidelines, 20-40% of the patients would need therapeutic intervention. For seizures longer than 3-5 minutes application of rectal diazepam, buccal midazolam or sublingual lorazepam is recommended. Benzodiazepines may be ineffective in some patients or cause prolonged sedation and fatigue. Preclinical investigations in a rat model provided evidence that febrile seizures may be triggered by respiratory alkalosis, which was subsequently confirmed by a retrospective clinical observation. Further, individual therapeutic interventions demonstrated that a pCO2-elevation via re-breathing or inhalation of 5% CO2 instantly stopped the febrile seizures. Here, we present the protocol for an interventional clinical trial to test the hypothesis that the application of 5% CO2 is effective and safe to suppress febrile seizures in children.

METHODS: The CARDIF (CARbon DIoxide against Febrile seizures) trial is a monocentric, prospective, double-blind, placebo-controlled, randomized study. A total of 288 patients with a life history of at least one febrile seizure will be randomized to receive either carbogen (5% CO2 plus 95% O2) or placebo (100% O2). As recurrences of febrile seizures mainly occur at home, the study medication will be administered by the parents through a low-pressure can fitted with a respiratory mask. The primary outcome measure is the efficacy of carbogen to interrupt febrile seizures. As secondary outcome parameters we assess safety, practicability to use the can, quality of life, contentedness, anxiousness and mobility of the parents.

PROSPECT: The CARDIF trial has the potential to develop a new therapy for the suppression of febrile seizures by redressing the normal physiological state. This would offer an alternative to the currently suggested treatment with benzodiazepines. This study is an example of academic translational research from the study of animal physiology to a new therapy.

TRIAL REGISTRATION: ClinicalTrials.gov identifier: NCT01370044. DOI: 10.1186/1479-5876-11-157 PMCID: PMC3700755 PMID: 23806032 [Indexed for MEDLINE]

ELIGIBILITY:
Inclusion Criteria:

* condition after febrile seizure
* age 12 months to 5 years
* written informed consent

Exclusion Criteria:

* severe other organic disease
* meningitis as possible cause for the cerebral seizure
* neurologic disease or cerebral dysplasia
* cerebrale seizures without fever in the medical history
* hypersynchronic eeg activity
* disorder of the respiratory tract (Asthma e.g.)

Ages: 12 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2012-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
number of patients which need Diazepam | 3 minutes
  efficacy of a Carbogen inhalation in patients with febrile seizures compared to a placebo inhalation

SECONDARY OUTCOMES:
number of severe adverse events | 3 minutes
  safety of the Carbogen inhalation via a low-pressure can with a breathing mask in a home-setting
manageability of the application assessed by the parents | 3 minutes
  manageability of the Carbogen inhalation via a low pressure can with a breathing mask in a home-setting or on the way (mobility)
changes in quality of life of the parents and children after use of study medication | 3 minutes
  quality of life of the parents and children using the low pressure can with a breathing mask in a home-setting or on the way (mobility)
contentment and anxiety of the parents | 10 minutes
  structured interview of the parents after a seizure

CONTACTS AND LOCATIONS:
Overall Officials: Markus Schülke-Gerstenfeld, Principal Investigator — Charite - NeuroCure
Locations (1):
- Charite University Berlin, Berlin, Germany

REFERENCES:
- [Background] Ohlraun S, Wollersheim T, Weiss C, Martus P, Weber-Carstens S, Schmitz D, Schuelke M. CARbon DIoxide for the treatment of Febrile seizures: rationale, feasibility, and design of the CARDIF-study. J Transl Med. 2013 Jun 27;11:157. doi: 10.1186/1479-5876-11-157. PMID 23806032
- [Derived] Weiss C, Hucko A, Muller-Ohlraun S, Marschenz S, Martus P, Schmitz D, Schuelke M. The use of carbogen for interruption of febrile seizures - the randomized controlled CARDIF trial. PLoS One. 2025 Dec 23;20(12):e0324422. doi: 10.1371/journal.pone.0324422. eCollection 2025. PMID 41433250
- See also: Homepage of the NeuroCure Clinical Resaerch Center at the Charité Berlin — https://neurocure.de/ncrc/ueber-uns.html